CLINICAL TRIAL: NCT03155711
Title: Study Protocol for the Use of High Flow Nasal Oxygen During the Anesthesia Induction and Weaning in Patients Scheduled for Bariatric Surgery. A Randomized Pilot Study
Brief Title: HFNC for Induction During Bariatric Surgery Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Carlos Ferrando, Principal Investigador, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HFNC-Obese
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Lung Collapse
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC (Experimental): HFNC with a 60 liters per minute flow will be given to the patients before anesthesia induction and before extubation at the end of the surgery
  Interventions: Procedure: HFNC group
- Standard (Active Comparator): This patients will be managed as usual care. Pre-oxygenation before induction will be performed with supplemental oxygen but without positive pressure. After extubation patients will be oxygenated through a ventury mask.
  Interventions: Procedure: Standard group

INTERVENTIONS:
Procedure: HFNC group — Positive pressure plus supplemental oxygen through a high flow nasal oxygen device
  Arms: HFNC
Procedure: Standard group — Supplemental oxygen through venturi mask
  Arms: Standard

SUMMARY:
This study aims to compared the effects of high flow nasal during the induction and during the weaning of anesthesia on intraoperative and postoperative oxygenation and postoperative atelectasis in obese patients undergoing bariatric surgery versus the standard of care, which consists in supplemental oxygen with face mask (Venturi mask).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index > 35 Kg/m2
* Bariatric surgery
* Informed consent signed

Exclusion Criteria:

* age <18yr or >80yr
* pregnancy or breast-feeding status
* patients with previous known respiratory disease
* hemodynamic instability at entry (need of vasopressors or ionotropes at entry or a ventricular assist device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Oxygenation | intraoperative
  The oxygenation (the ratio of partial pressure of arterial oxygen with inspiratory oxygen fraction, PaO2/FIO2) informs of the percentadge of shunt.

SECONDARY OUTCOMES:
Oxygenation | First 24 postoperative hours
  PaO2/FIO2
Atelectasis | First 24 postoperative hours
  Atelectasis evaluated with X-ray

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital clínico universitario, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eichenberger A, Proietti S, Wicky S, Frascarolo P, Suter M, Spahn DR, Magnusson L. Morbid obesity and postoperative pulmonary atelectasis: an underestimated problem. Anesth Analg. 2002 Dec;95(6):1788-92, table of contents. doi: 10.1097/00000539-200212000-00060. PMID 12456460
- [Background] Coussa M, Proietti S, Schnyder P, Frascarolo P, Suter M, Spahn DR, Magnusson L. Prevention of atelectasis formation during the induction of general anesthesia in morbidly obese patients. Anesth Analg. 2004 May;98(5):1491-5, table of contents. doi: 10.1213/01.ane.0000111743.61132.99. PMID 15105237
- [Background] Ireland CJ, Chapman TM, Mathew SF, Herbison GP, Zacharias M. Continuous positive airway pressure (CPAP) during the postoperative period for prevention of postoperative morbidity and mortality following major abdominal surgery. Cochrane Database Syst Rev. 2014 Aug 1;2014(8):CD008930. doi: 10.1002/14651858.CD008930.pub2. PMID 25081420